CLINICAL TRIAL: NCT03250858
Title: Randomized Control Trial to Evaluate the Effectiveness of Online Nutrition Advice in the UK (The EatWellUK Study)
Brief Title: Online Nutrition Advice in the UK (EatWellUK)
Acronym: EatWellUK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13/17
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Dietary Modification; Dietary Habits
Keywords: Personalised nutrition; Mobile web application
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-personalised advice (Placebo Comparator): Control group. Online (web-based) delivery of non-personalised dietary, weight and physical activity advice based on the UK general health guidelines.
  This is an online trial and this arm will be using the e-Nutri web application. Participants in this group will receive online general recommendations (non-personalised).
  Interventions: Behavioral: Non-personalised advice
- Personalised advice (Experimental): Online (web-based) delivery of personalised dietary, weight and physical activity advice based on the individual's dietary intake, weight and physical activity levels, generated by the e-Nutri web application. Participants in this group will receive online personalised reports.
  Interventions: Behavioral: Personalised advice

INTERVENTIONS:
Behavioral: Personalised advice — Provision of online personalised advice on dietary intake, weight and physical activity levels. Personalised recommendations for improved food choice based on adherence to an 11-item modified US Alternative Healthy Eating Index (m-AHEI), for weight based on ideal BMI range and for physical activity based on the Baecke questionnaire/results.
  Arms: Personalised advice
Behavioral: Non-personalised advice — Provision of online non-personalised advice on dietary intake, weight and physical activity levels. Non-personalized dietary advice for improved food choice based on standard population health guidelines.
  Arms: Non-personalised advice

SUMMARY:
The EatWellUK study aims to investigate the effectiveness of a mobile web application (e-Nutri), capable of delivering automated personalised nutrition advice, in increasing diet quality.

Dietary assessment is via the validated Food4Me FFQ (with an updated user interface that has been designed for better usability) and dietary feedback is derived according to adherence to an 11-item modified US Alternative Healthy Eating Index (m-AHEI).

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years old

Exclusion Criteria:

* aged < 18 years old
* not living in the UK
* pregnant/lactating
* no or limited access to internet
* following a prescribed diet for any reason
* intolerance or food allergy
* subject with diabetes, or any other metabolic disorder or illness that alters nutritional requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Dietary intake | baseline, 6 weeks, 12 weeks
  Change from baseline in dietary intake at 6 and 12 weeks assessed via a Food Frequency Questionnaire (FFQ). An 11-item modified US Alternative Healthy Eating Index (m-AHEI), which is calculated from the results of the FFQ, will be used to quantify the dietary intake changes.

SECONDARY OUTCOMES:
Weight | baseline, 6 weeks, 12 weeks
  Change from baseline in self-reported weight (kg) at 6 and 12 weeks. Weight variation will be combined with height (constant for adults) and also reported as BMI variation (kg/mˆ2).
Physical activity | baseline, 6 weeks, 12 weeks
  Change from baseline in self-reported physical activity (Baecke questionnaire) at 6 and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Zenun Franco R, Fallaize R, Weech M, Hwang F, Lovegrove JA. Effectiveness of Web-Based Personalized Nutrition Advice for Adults Using the eNutri Web App: Evidence From the EatWellUK Randomized Controlled Trial. J Med Internet Res. 2022 Apr 25;24(4):e29088. doi: 10.2196/29088. PMID 35468093